CLINICAL TRIAL: NCT00937508
Title: A Double Blind Randomized Placebo Controlled Study, for Smoking Cessation in Preadmission Clinic. the Use of a Teachable Moment
Brief Title: Smoking Cessation Program in the Preadmission Clinic
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Dr. Frances Chung, Anesthesia Department, Toronto Western Hospital, University Health Network
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-0585-AE; Protocol# in Pfizer: GA30517W
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Last update posted 2010-04-08 (Estimated); Status verified 2010-01

CONDITIONS: Smoking
Keywords: smoking; quitting; varenicline; preoperative; long term abstinence
MeSH Terms: conditions — Smoking | interventions — Counseling; Varenicline; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Smoking counseling, Placebo (Placebo Comparator)
  Interventions: Behavioral: Smoking counseling; Drug: placebo
- Smoking counseling, Varenicline (Experimental)
  Interventions: Behavioral: Smoking counseling; Drug: varenicline

INTERVENTIONS:
Behavioral: Smoking counseling — Preoperative and postoperative counseling sessions provided by a trained smoking counselor along with placebo.
  Other Names: counseling for smoking cessation
Drug: varenicline — varenicline (an approved medication for smoking cessation)
  Other Names: Champix, Chanitx
  Arms: Smoking counseling, Varenicline
Drug: placebo — sugar pill without any active medication
  Other Names: sugar pill (control)
  Arms: Smoking counseling, Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled clinical trial which evaluates the efficacy of preoperative smoking counseling and varenicline (a medication approved by Health Canada and FDA for quitting smoking) to provide long term smoking cessation (i.e., abstinence for at least one year) in surgical patients.

The primary hypothesis is as follows: "A significant percentage of surgical patients will be receptive to smoking cessation interventions in the pre-admission clinic and will refrain from smoking at 24 and 52 weeks after starting the treatment." The secondary hypothesis is as follows: "Patients who receive interventions but do not quit smoking will have reduced number of cigarettes consumed/day or improved their readiness to quit smoking at 24 and 52 weeks after starting the treatment."

DETAILED DESCRIPTION:
The Objective of this study is to introduce a practically feasible multifaceted intervention in the preadmission clinic to help reduce smoking in preoperative surgical patients. We aim to study the effectiveness of such a program in promoting positive change in smoking behavior among patients before surgery. The forced abstinence enforced on patients during hospital stay for their surgery can also be used to help smokers remain tobacco free long term.

The intervention program for this study will be primarily based on the smoking cessation guidelines endorsed by the Department of Family and Community Medicine, University of Toronto. The study research staffs (including the research coordinator) will be trained in accordance with these guidelines and the reading material provided will also be based on the same guidelines. The counseling skills of the coordinator will be reviewed every 3 months to ensure minimal variability. The coordinator will also be involved in regular meetings to address difficult situations and scenarios. They will also be provided checklists for all interventions to ensure that all components are covered uniformly for each patient. For each patient, the research staff who interviews the patient at the beginning will be the same during the whole treatment and follow-up period.

Interventions in Preadmission:

Demographic and personal chrematistics of the patients including age, sex, average number of cigarette smoked per day will be recorded. Patients will then receive a questionnaire based on Prochaska and DiClemente's Stages of Change Model to determine whether they were precontemplating, contemplating, preparing for or actively engaged in smoking cessation. In order to have the baseline smoking status, urinary cotinine and expired-air carbon monoxide (COE) will be measured in all patients at the preadmission clinic.

All patients will receive two 15 minute face to face standard counseling sessions by the research coordinator. First counseling will be done in preadmission. Counseling will include provision of advice to quit smoking and obtaining information regarding smoking behavior and skill building supplemented with standard printed materials. The patients will be informed of benefits of even short term abstinence before surgery. The target quit date (TQD) for all patients will be set up as 24 hours before surgery as surgical patients are routinely required to be abstinent at the time of surgery. The patients will be instructed to initiate the medication (or placebo) exactly one week before TQD. The whole treatment period is 12 weeks which includes 1- week titration as follows:

Days 1 - 3: 0.5 mg once daily (1 table each day) Days 4 - 7: 0.5 mg twice daily (1 in the morning and 1 in the evening) Days 8 - 12 weeks 1.0 mg twice daily (1 in the morning and 1 in the evening)

Patients in the varenicline group will be prescribed varenicline for 12 weeks. Patients in the placebo group will be prescribed placebo (lactose, identical to medication pills in appearance) for the same period of time.

The patients at the preadmission clinic will receive two bottles of the medication (or placebo): One containing 17 X 0.5 mg tabs (i.e. 11 tabs plus 6 extra tablets for a 3-day window period) for the first week of titration; the other one containing 66 X 1.0 mg tabs (28 days X 2 tablets = 56 tablets plus10 for a 5-day window period) for the next 4 weeks of treatment. We will call the patients one week before TQD to remind them to start the treatment. In case of delayed or cancelled surgeries, TQD will not change and the patient will continue the treatment according to the above mentioned schedule. The patients will be asked to return the first medication bottle with the remaining pills on the day of surgery.

There have been rare post-marketing reports of serious neuropsychiatric symptoms with varenicline, including depressed mood, agitation, hostility, changes in behavior, suicidal ideation and suicide, as well as worsening of pre-existing psychiatric illness (previously diagnosed or not). It is not known whether these events are occurring at a rate and severity which is different from the background rate for smoking cessation in the general population, or in the psychiatric population (treated or untreated), or different from the rates for other drugs in the class of smoking cessation.

All patients and/or their families will be alerted about the need to monitor for the medication side effects including any neuropsychiatric symptoms. Since the beginning of the treatment and during each in-hospital visit or follow up phone calls, patients will be asked about changes in their behavior or thoughts. Patients will be instructed to stop taking the medication (or placebo) and contact their healthcare provider and the research coordinator immediately if they have or if their families observe depressed mood, agitation, hostility or changes in behavior, that are not typical for the patient, or if the patient has suicidal ideation or suicidal behavior. These patients will be unblinded, withdrawn from the study, and recorded as cases with serious adverse events (SAE). They will be followed up for at least 28 days after the stop of the treatments for monitoring any more complications.

Intervention during hospital admission:

On the day of surgery, the patients will take one pill of 1.0 mg medication (or matched placebo) before surgery. They will resume taking the medication as soon as possible after surgery according to the treatment schedule. At 24 hour after surgery or discharge time (for day-surgery patients), i.e. the postoperative visit, patients will receive the rest of medications for the whole treatment period, i.e. two bottles of the medication (or placebo) each one containing 66 X 1.0 mg tabs (28 days X 2 tablets = 56 tablets plus10 for a 5-day window) for the rest of treatment.

Any interruption in the treatment which might happen due to patient surgical conditions (e.g. patients having abdominal surgeries, etc.) will be recorded for taking into account in the final sub-analysis. The second counseling session will be at discharge for day-surgery patients or at 24 hrs after other surgeries. Participants will be visited by the study coordinator in the hospital to review smoking status and to encourage future abstinence. The self-reported preoperative abstinence will then be verified by measurement of expired carbon monoxide (COE) and urinary cotinine in all patients. Patients will receive counseling with special emphasis on the skills associated with relapse prevention and remaining abstinent during second week as research suggests that abstinence during that time period is highly predictive of success (Kenford et al 1994) and promotes surgical healing (Warner et al 2004). Patients will also be informed of benefits of long-term cessation and will be encouraged to continue pharmacotherapy.

Long-term follow up and telephone counseling after discharge:

Participants in both groups will also be provided with telephone counseling. For the first 4 weeks after starting treatment, the patients will receive weekly phone calls and then at the end of 8 weeks. The purpose of these calls will be to report smoking status and to help encourage continued and long-term abstinence. Patients then will be asked to come to the hospital for a visit at the end of their treatment period, i.e. 12 weeks after the treatment started. They will be compensated for the traveling and parking cost and required to bring the bottles including the remaining pills. In this visit, patients will be asked about their smoking status and their stage of change using Prochaska and DiClemente's model or no. of cigarette smoked/ day for those who have not quit smoking. In addition, the self-reported abstinence will then be verified by measurement of expired carbon monoxide (COE) and urinary cotinine in all patients. For the rest of follow-up period, i.e. until the end of week 52 after treatment, patients will receive phone calls every 4 weeks to encourage continued and long-term abstinence. The smoking status, stage of change and no. of cigarette smoked/ day will also be reported at 24- and 52- week follow-up phone calls. To verify self-reports of abstinence, we will also mail the NicAlert urine cotinine strips (Accutest) at 24 and 52 weeks after treatment to the patients along with instructions of how to do the test. Patients will be asked by telephone calls to do the test and to return the strips using prepaid return envelops including a small plastic pouch.

Patients will be followed up for 52 weeks after starting the treatment. Participants in both groups will receive a follow up visit by the study coordinator or a research assistant during their hospital stay i.e., at discharge for day surgery patients or at 24 hrs after their surgery. Patients in both groups will receive weekly follow up calls during the first 4 weeks and then at the end of 8 week after starting the treatment. At the end of treatment period, i.e. 12 weeks patients will come be visited in the hospital. For the rest of follow-up period, i.e. until the end of week 52, patients will receive phone calls for every 4 weeks to help support abstinence and to report smoking status. Focus will be on the second week following start of abstinence as it has been shown that abstinence of smoking at 2 wks after a cessation attempt is highly predictive of success. The self reports of smoking status at 24- and 52-week follow-up will be verified by measuring COE and urine cotinine.

ELIGIBILITY:
Inclusion Criteria:

* patients who are assessed in pre-admission clinic and scheduled for elective surgical procedures within the next 8 to 30 days
* patients should be over 18 yrs of age
* patients should have smoked an average 10 cigarettes/day or more during the previous year and had no period of smoking abstinence longer than 3 months in the past year

Exclusion Criteria:

* current pregnancy (or willingness to be pregnant within the next year after the start of the medication)
* current breastfeeding
* major depression, panic disorder, psychosis, or bipolar disorder within the prior year
* use of nicotine replacement or bupropion within the previous 3 months cardiovascular disease within the past 6 months
* a serious or unstable disease within the past 6 months
* drug or alcohol abuse or dependence within the past year
* use of tobacco products other than cigarettes or marijuana use within the previous month
* participating in any other studies
* patients who cannot understand English or have any form of cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-07 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Point prevalence of smoking cessation (those who have quitted smoking and have not smoked in the past week prior to the assessment date). | 52 weeks after starting the treatment

SECONDARY OUTCOMES:
Point prevalence of smoking cessation (those who have quitted smoking and have not smoked in the past week prior to the assessment date). | 24 weeks after starting the treatment.
Number of cigarettes consumed per day over the past week prior to the assessment date. | 52 weeks after starting the treatment
Number of cigarettes consumed per day over the past week prior to the assessment date. | 24 weeks after starting the treatment
"stage of change" (determined by Prochaska and DiClemente's Model) | 52 weeks after starting the treatment
Total prevalence of drug-related adverse events | after treatment unitl one month after the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Frances Chung, FRCPC, Principal Investigator — Anesthesia Department, Toronto Western Hospital, University of Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Streck JM, Rigotti NA, Livingstone-Banks J, Tindle HA, Clair C, Munafo MR, Sterling-Maisel C, Hartmann-Boyce J. Interventions for smoking cessation in hospitalised patients. Cochrane Database Syst Rev. 2024 May 21;5(5):CD001837. doi: 10.1002/14651858.CD001837.pub4. PMID 38770804
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273